CLINICAL TRIAL: NCT03853018
Title: The Effectiveness of Consumer Wearable Activity Trackers to Reduce Sedentary Behaviour and Improve Health-related Outcomes in Sedentary Adults
Brief Title: Effectiveness of Activity Trackers to Reduce Sedentary Behaviour in Sedentary Adults
Acronym: CWATLDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Bert Op't Eijnde, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CWATLDP-001
Record Dates: First submitted 2018-11-15; First posted 2019-02-25 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): The control group is instructed to continue their habitual daily physical activity patterns and sedentary behaviour
- CWAT intervention group (Experimental): The CWAT group will receive the activity tracker. Subjects will receive inactivity alerts after 1 hour of inactivity to break up sitting time and avoid prolonged sitting. During the interruptions they will be asked to walk for several minutes.
  Interventions: Device: CWAT intervention
- CWAT + motivation intervention group (Experimental): Subjects randomised into the CWATLDP intervention will receive the activity tracker and will be stimulated with the aid of coaching sessions and goal setting.
  Interventions: Device: CWAT intervention; Device: CWAT + motivation intervention group

INTERVENTIONS:
Device: CWAT intervention — Participant in the intervention group will wear an activity tracker for 12 weeks.
  Arms: CWAT + motivation intervention group; CWAT intervention group
Device: CWAT + motivation intervention group — Participant in the intervention group will wear an activity tracker for 12 weeks and are also motivated by the researcher via a lifestyle data platform.
  Arms: CWAT + motivation intervention group

SUMMARY:
This study evaluates the effectiveness of consumer wearable activity trackers to reduce sedentary behaviour and the impact on cardiometabolic health.

DETAILED DESCRIPTION:
Chronic non-communicable diseases (NCDs), including cardiovascular diseases, cancer, chronic respiratory diseases and diabetes, are an important public health concern worldwide. Physical inactivity is one of the major contributing factors which is highly correlated with the prevalence of NCDs. On the other hand, it is well known that increased physical activity has significant health benefits and is associated with the prevention and delayed onset of many NCDs. Given the important role of physical activity in the prevention and management of NCDs it is thus important to promote physical activity. Hence, to date a multitude of physical activity recommendations and many supervised training interventions and rehabilitation programs are available to encourage physical activity in the global population. Despite this, a recent report from the World Health Organization (WHO) indicates that 23% of the adult and 80% of the adolescent population remains physically inactive. Here, long-term compliance to adequate physical activity and a healthy life style appears to be one of the main barriers explaining this discrepancy. Consequently, any strategy that improves long term adherence to adequate daily physical activity and a healthy life style, especially in an NCD population, is worthwhile investigating. In this respect and following the recent use of accelerometer-based remote monitoring of physical activity in chronic disease patients, consumer wearable activity trackers may be such a strategy. So far, consumer wearable activity trackers have been investigated mainly in the sports community. Here CWATs are used for self-monitoring and providing continuous sport performance and health related information to athletes and coaches. Interestingly, the self-management, motivational and goal setting properties of these commercially available devices may also help patients with NCDs to engage in long-term physical activity under free-living conditions in a home-based setting. Despite the widespread use of these wearables their feasibility and effectiveness on physical activity (compliance) and generic health-related outcomes, including weight, body mass index (BMI), systemic blood pressure and glycemic index, especially in patients with NCDs is not fully clear.

Therefore, the aim of this study is to investigate the effectiveness of CWATs to promote physical activity levels and cardiometabolic health in sedentary adults. A better understanding to what extent CWATs can actually improve physical activity (compliance) and health outcomes is important to increase the effectiveness and quality of health care in chronic disease populations.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary adults
* 40-75 years,
* <7500steps/day,
* sitting time of >10h/day,
* BMI 23-30 kg/m2,
* body fat percentage: male: 18-25%, female: 25-35%
* HbA1c < 6.0%

Exclusion Criteria:

* pregnancy,
* regularly (>150 min per week during the last four months) engaged in moderate-to-vigorous intensity exercise,
* any known contradiction for physical activity,
* systolic blood pressure >160mmHg,
* diastolic blood pressure >100mmHg
* more than 20 alcohol consumptions per week,
* plans to follow a weight reduction program with the aid of an energy restriction diet or a physical intervention program during the study period,
* participants diagnosed with any known chronic disease.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Steps per day | Baseline
  Physical activity will be quantified using the activPAL3™ activity monitor.
sitting time | baseline
  sedentary behaviour will be quantified using the activPAL3™ activity monitor.
Steps per day | week 12
  Physical activity will be quantified using the activPAL3™ activity monitor.
sitting time | week 12
  sedentary behaviour will be quantified using the activPAL3™ activity monitor.

SECONDARY OUTCOMES:
body weight | baseline
  Body weight (in underwear) is determined using a digital-balanced weighting scale to the nearest 0.1kg
body weight | week 12
  Body weight (in underwear) is determined using a digital-balanced weighting scale to the nearest 0.1kg
Height | baseline
  Body height is measured to the nearest 0.1cm using a wall-mounted Harpenden stadiometer, with participants barefoot
Height | week 12
  Body height is measured to the nearest 0.1cm using a wall-mounted Harpenden stadiometer, with participants barefoot
DEXA (Dual Energy X-Ray) | baseline
  body fat mass and lean tissue mass using Dual Energy X-ray Absorptiometry
DEXA (Dual Energy X-Ray) | week 12
  body fat mass and lean tissue mass using Dual Energy X-ray Absorptiometry
Concentration of glucose | baseline
  Blood analysis
Concentration of glucose | week 12
  Blood analysis
Concentration of Insuline | baseline
  Blood analysis
Concentration of Insuline | week 12
  Blood analysis
Concentration of total cholesterol | baseline
  Blood analysis
total cholesterol | week 12
  Blood analysis
Concentration of high density lipoprotein cholesterol (HDL-cholesterol) | baseline
  Blood analysis
Concentration of high density lipoprotein cholesterol (HDL-cholesterol) | week 12
  Blood analysis
Concentration of low density lipoprotein cholesterol (LDL-cholesterol) | baseline
  Blood analysis
Concentration of low density lipoprotein cholesterol (LDL-cholesterol) | week 12
  Blood analysis
Concentration of triglyceride | baseline
  Blood analysis
Concentration of triglyceride | week 12
  Blood analysis
Concentration of glycated haemoglobin (HbA1c) | baseline
  Blood analysis
Concentration of glycated haemoglobin (HbA1c) | week 12
  Blood analysis
Concentration of uric acid | baseline
  Blood analysis
Concentration of uric acid | week 12
  Blood analysis
Concentration of interleukin 6 (IL-6), | baseline
  Blood analysis
Concentration of interleukin 6 (IL-6), | week 12
  Blood analysis
Concentration of tumor necrosis factor-alpha (TNF-α), | baseline
  Blood analysis
Concentration of tumor necrosis factor-alpha (TNF-α), | week 12
  Blood analysis
Concentration of C-reactive protein (CRP) | baseline
  Blood analysis
Concentration of C-reactive protein (CRP) | week 12
  Blood analysis
Concentration of serum amyloid A (SAA) | baseline
  Blood analysis
Concentration of serum amyloid A (SAA) | week 12
  Blood analysis
Concentration of soluble vascular cell adhesion molecule-1 (sVCAM-1), | baseline
  Blood analysis
Concentration of soluble vascular cell adhesion molecule-1 (sVCAM-1), | week 12
  Blood analysis
Concentration of soluble intercellular adhesion molecule 1 (sICAM-1) | baseline
  Blood analysis
Concentration of soluble intercellular adhesion molecule 1 (sICAM-1) | week 12
  Blood analysis
Concentration of soluble E-selectin (sE-selectin). | baseline
  Blood analysis
Concentration of soluble E-selectin (sE-selectin). | week 12
  Blood analysis
Vascular endothelial function | baseline
  Endothelial function will be assessed by non-invasive peripheral arterial tonometry using the EndoPAT™ 2000 device
Vascular endothelial function | week 12
  Endothelial function will be assessed by non-invasive peripheral arterial tonometry using the EndoPAT™ 2000 device
Homeostatic model assessment for insulin resistance (HOMA-IR) | baseline
  An oral glucose tolerance test will be performed for assessment of whole body insulin sensitivity using the homeostatic model assessment for insulin resistance (HOMA-IR). The HOMA-IR is calculated from the fasting insulin and glucose concentration.sensitivity and beta cell function. The following parameters are calculated: homeostatic model assessment for insulin resistance, whole-body insulin sensitivity index, insulinogenic index and the area under the curve for glucose and insulin.
Homeostatic model assessment for insulin resistance (HOMA-IR) | week 12
  An oral glucose tolerance test will be performed for assessment of whole body insulin sensitivity using the homeostatic model assessment for insulin resistance (HOMA-IR). The HOMA-IR is calculated from the fasting insulin and glucose concentration.sensitivity and beta cell function. The following parameters are calculated: homeostatic model assessment for insulin resistance, whole-body insulin sensitivity index, insulinogenic index and the area under the curve for glucose and insulin.
Whole-body insulin sensitivity index (ISI) | baseline
  An oral glucose tolerance test will be performed for assessment of whole body insulin sensitivity using the whole-body insulin sensitivity index (ISI). The ISI is calculated from both insulin and glucose concentrations.
Whole-body insulin sensitivity index (ISI) | week 12
  An oral glucose tolerance test will be performed for assessment of whole body insulin sensitivity using the whole-body insulin sensitivity index (ISI). The ISI is calculated from both insulin and glucose concentrations.
Area under the curve of insulin concentrations | baseline
  An oral glucose tolerance test will be performed for assessment of whole body insulin sensitivity by calculation of the area under the curve of insulin concentrations.
Area under the curve of insulin concentrations | week 12
  An oral glucose tolerance test will be performed for assessment of whole body insulin sensitivity by calculation of the area under the curve of insulin concentrations.
Area under the curve of glucose concentrations | baseline
  An oral glucose tolerance test will be performed for assessment of whole body insulin sensitivity by calculation of the area under the curve of glucose concentrations.
Area under the curve of glucose concentrations | week 12
  An oral glucose tolerance test will be performed for assessment of whole body insulin sensitivity by calculation of the area under the curve of glucose concentrations.
Insulinogenic index | baseline
  An oral glucose tolerance test will be performed for assessment of beta cell function by calculation of the insulinogenic index. The insulinogenic index is calculated from both insulin and glucose concentrations.
Insulinogenic index | week 12
  An oral glucose tolerance test will be performed for assessment of beta cell function by calculation of the insulinogenic index. The insulinogenic index is calculated from both insulin and glucose concentrations.
Cardiac autonomic function | baseline
  Cardiac autonomic function will be operationalized as heart rate variability by means of continuous beat-to-beat heart rate signal measurements. time domain and frequency domain analysis of the R-R intervals will be performed
Cardiac autonomic function | week 12
  Cardiac autonomic function will be operationalized as heart rate variability by means of continuous beat-to-beat heart rate signal measurements. time domain and frequency domain analysis of the R-R intervals will be performed
Systolic and Diastolic Blood pressure | baseline
  Systolic, diastolic and mean arterial blood pressure will be measured 3 times at 5-min intervals using an electronic sphygmomanometer
Systolic and Diastolic Blood pressure | week 12
  Systolic, diastolic and mean arterial blood pressure will be measured 3 times at 5-min intervals using an electronic sphygmomanometer
Oxygen uptake (VO2) | baseline
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VO2 is collected breath-by-breath and averaged every ten seconds.
Oxygen uptake (VO2) | week 12
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VO2 is collected breath-by-breath and averaged every ten seconds.
Carbon dioxide output (VCO2) | baseline
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VCO2 is collected breath-by-breath and averaged every ten seconds.
Carbon dioxide output (VCO2) | week 12
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VCO2 is collected breath-by-breath and averaged every ten seconds.
Minute ventilation (VE) | baseline
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VE is collected breath-by-breath and averaged every ten seconds.
Minute ventilation (VE) | week 12
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VE is collected breath-by-breath and averaged every ten seconds.
Equivalents for oxygen uptake (VE/VO2) | baseline
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VE/VO2 is collected breath-by-breath and averaged every ten seconds.
Equivalents for oxygen uptake (VE/VO2) | week 12
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VE/VO2 is collected breath-by-breath and averaged every ten seconds.
Equivalents for carbon dioxide production (VE/VCO2) | baseline
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VE/VCO2 is collected breath-by-breath and averaged every ten seconds.
Equivalents for carbon dioxide production (VE/VCO2) | week 12
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VE/VCO2 is collected breath-by-breath and averaged every ten seconds.
Tidal volume (Vt) | baseline
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis Vt is collected breath-by-breath and averaged every ten seconds.
Tidal volume (Vt) | week 12
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis Vt is collected breath-by-breath and averaged every ten seconds.
Breathing frequency (BF) | baseline
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis BF is collected breath-by-breath and averaged every ten seconds.
Breathing frequency (BF) | week 12
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis BF is collected breath-by-breath and averaged every ten seconds.
Respiratory gas exchange ratio (RER) | baseline
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis RER is collected breath-by-breath and averaged every ten seconds.
Respiratory gas exchange ratio (RER) | week 12
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis RER is collected breath-by-breath and averaged every ten seconds.
Heart rate (HR) | baseline
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of a heart rate monitor the HR is measured and averaged every ten seconds.
Heart rate (HR) | week 12
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of a heart rate monitor the HR is measured and averaged every ten seconds.
A six-minute walk test | baseline
  The covered distance is measured during a six-minute walk test.
A six-minute walk test | week 12
  The covered distance is measured during a six-minute walk test.
Relative autonomy index | baseline
  Individual motives for physical activity are assessed using the Behavioural Regulation and Exercise Questionnaire version 2 (BREQ-2).
Relative autonomy index | week 12
  Individual motives for physical activity are assessed using the Behavioural Regulation and Exercise Questionnaire version 2 (BREQ-2).
Total calorie intake | baseline
  Participants will record all food and beverages consumed over seven consecutive days and from this the total calorie intake is calculated.
Total calorie intake | week 12
  Participants will record all food and beverages consumed over seven consecutive days and from this the total calorie intake is calculated.
Macronutrient content | baseline
  Participants will record all food and beverages consumed over seven consecutive days and from this the macronutrient content is calculated.
Macronutrient content | week 12
  Participants will record all food and beverages consumed over seven consecutive days and from this the macronutrient content is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Bert Op 't Eijnde, prof. dr., Study Chair — Hasselt University; Wouter Franssen, drs., Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Diepenbeek, Limburg, Belgium

REFERENCES:
- [Derived] Franssen WMA, Nieste I, Vandereyt F, Savelberg HHCM, Eijnde BO. A 12-week consumer wearable activity tracker-based intervention reduces sedentary behaviour and improves cardiometabolic health in free-living sedentary adults: a randomised controlled trial. J Act Sedentary Sleep Behav. 2022 Dec 1;1(1):8. doi: 10.1186/s44167-022-00007-z. PMID 40229981